CLINICAL TRIAL: NCT07047703
Title: A Multi-part, Phase I/II Study to Evaluate the Safety and Tolerability of GRWD0715 in Healthy Human Volunteers and Participants With Axial Spondyloarthritis
Brief Title: EAST-1 (ERAP-inhibition in Axial Spondyloarthritis Trial - 1)
Acronym: EAST-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grey Wolf Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GRWD0715-AS-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Axial Spondyloarthritis (AxSpA)
Keywords: Axial Spondyloarthritis; AxSpA
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Masking Description: Parts A, B, and C - None (Open Label). Part D will be double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A - Single Ascending Dose (SAD) in Healthy Human Volunteers (Experimental)
  Interventions: Drug: Part A - Single Ascending Dose (SAD) in Healthy Human Volunteers
- Part B - Multiple Ascending Dose (MAD) in participants with axSpA (Experimental)
  Interventions: Drug: Part B - Multiple Ascending Dose (MAD) in participants with axSpA
- Part C - Safety expansion cohort in participants with axSpA (Experimental)
  Interventions: Drug: Part C - Safety expansion cohort in participants with axSpA
- Part D - Randomised, placebo-controlled, expansion cohort in participants with axSpA (Experimental)
  Interventions: Drug: Part D - Randomised, placebo-controlled, expansion cohort in participants with axSpA

INTERVENTIONS:
Drug: Part A - Single Ascending Dose (SAD) in Healthy Human Volunteers — Participants in Part A will receive a single dose of GRWD0715 on Day 1 only.
  Arms: Part A - Single Ascending Dose (SAD) in Healthy Human Volunteers
Drug: Part B - Multiple Ascending Dose (MAD) in participants with axSpA — Participants in Part B will receive GRWD0715 for 28 days
  Arms: Part B - Multiple Ascending Dose (MAD) in participants with axSpA
Drug: Part C - Safety expansion cohort in participants with axSpA — Participants in Part C will receive GRWD0715 for 12 weeks
  Arms: Part C - Safety expansion cohort in participants with axSpA
Drug: Part D - Randomised, placebo-controlled, expansion cohort in participants with axSpA — Participants in Part D will receive GRWD0715 or placebo-to-match for 12 weeks
  Arms: Part D - Randomised, placebo-controlled, expansion cohort in participants with axSpA

SUMMARY:
GRWD0715 is an orally administered, selective inhibitor of the Endoplasmic Reticulum Aminopeptidase 1 [ERAP1] enzyme being explored as a potential new treatment for axial spondyloarthritis (axSpA), a long term condition caused by inflammation predominantly affecting the sacroiliac joints (SIJs) and spine.

DETAILED DESCRIPTION:
GRWD0715 is an orally administered, selective inhibitor of the Endoplasmic Reticulum Aminopeptidase 1 [ERAP1] enzyme being explored as a potential new treatment for axial spondyloarthritis (axSpA), a long term condition caused by inflammation predominantly affecting the sacroiliac joints (SIJs) and spine.

ERAP1 is involved in trimming antigens from foreign bodies (e.g. bacteria, viruses) which are presented on the surface of a cell to trigger an immune response. In axSpA, it is thought an antigen from the person's own body, called a 'self-peptide' is presented by the ERAP1 processing pathway and incorrectly recognised by the immune system. The hypothesis is that stimulation of the immune system by the presentation of this self-peptide causes the inflammatory symptoms experienced by people living with axSpA.

As an inhibitor of ERAP1, GRWD0715 aims to prevent the generation of the antigenic self-peptide, and thus remove the stimulus of the immune system. If the immune system is not activated, the immune attack on the sacroiliac joint (SIJ) and spine would stop, halting the axSpA disease progress.

The study will consist of 4 parts: Part A conducted in healthy human volunteers, and Part B, Part C and/or D in participants with axSpA. The primary goal of Parts A, B and C is to assess whether GRWD0715 is safe and well tolerated in healthy human volunteers and participants with axSpA. The primary goal of Part D is to review whether GRWD0715 is efficacious when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* Healthy male and female subjects aged 18-55 years inclusive, at the Screening visit
* Participant must provide written informed consent to participate in the study
* Participant must be able and willing to comply with the requirements of the protocol (including dietary restrictions and exclusion of grapefruit juice)
* Male participants (and their female partners) / female participants must be willing to adhere to contraception requirements as detailed in the protocol
* Non-smokers or ex-smokers who have not smoked within the previous 6 months, as determined at the Screening visit
* Participant with a Body Mass Index (BMI) of 19-30. Body Mass Index = Body weight (kg) / [Height (m)]2

AxSpA Participants

* Male or female, 18-65 years of age
* Participants diagnosed with Axial Spondyloarthritis, also fulfilling ASAS classification criteria including:

  1. HLA-B27 +ve (local testing)
  2. Objective evidence of inflammation at screening, specifically active sacroiliac joint inflammation on MRI fulfilling the ASAS MRI criteria (MRI+), assessed by the Principal Investigator or appropriately trained delegate, and/or elevated C-reactive protein (CRP+) ≥5.0mg/L.
* Symptom duration of ≥3 months
* Age at onset of active disease of <40 years
* A score of ≥ 2.1 on the Ankylosing Spondylitis Disease Activity Score (ASDAS) on current treatment.
* At least one of the following:

  1. Current treatment with a NSAID, at a sufficient dose and following an appropriate dosing duration per local clinical guidelines, with inadequate clinical response OR
  2. Intolerance to ≥1 NSAID or contraindication(s) to NSAIDs
* Participants may have received 1 prior/(Australia only) 2 prior b/ts DMARD and discontinued due to intolerance or inadequate efficacy.
* Participants who have received 1/(Australia only) 2 prior treatments are required to undergo a washout at minimum:

  1. Biologic DMARDs 4 weeks or 5 half-lives prior to Day 1, whichever is longer.
  2. JAK inhibitor DMARDs 2 weeks prior to Day 1

Exclusion Criteria:

Healthy Volunteers

* History or presence of any clinically significant findings in medical history, physical examination, vital signs and/or laboratory tests that, in the opinion of the Investigator, would preclude inclusion in the study
* Participation in a New Chemical Entity clinical study within the previous 124 days or a marketed drug clinical study within the previous 93 days
* Known infection or lifestyle risk factors for human immunodeficiency virus (HIV) and/or hepatitis B or C infection, as determined at the Screening visit

AxSpA Participants

* Participants who have received >1/(Australia only) >2 biologic or JAK inhibitor DMARD or are receiving any other disease-modifying antirheumatic drugs (other than those allowed), thalidomide (including previous use) and other prohibited concomitant medications.
* Inadequate Haematologic function, defined as:

  1. Haemoglobin <10 g/dL.
  2. Absolute white blood cell count <3.0 x 109 /L (<3000 mm3)
  3. Absolute neutrophil count <1.2 x 109 /L (<1200 mm3)
  4. Absolute lymphocyte count <1.0 x 109 /L (<1000 mm3)
  5. Platelet count <100 x 109 /L (<100.000 mm3)
* Inadequate liver function, defined as; total bilirubin, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal at screening visit. For subjects with Gilberts syndrome, upper limit of normal for total bilirubin will be 2.9mg/dl
* History of any other autoimmune rheumatic disease (e.g., psoriatic arthropathy, systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymositis) or known diagnosis of fibromyalgia
* Participants with a previous history of or currently stable psoriasis are eligible
* Active or symptomatic inflammatory bowel disease (IBD). Participants with a history of IBD are allowed to participate
* Presence of active anterior uveitis

Please note the following Country-Specific Inclusion Criteria, for study participants in Australia:

- Participants with a score of ≥ 2.1 (High Disease Activity) on the Ankylosing Spondylitis Disease Activity Score (ASDAS) on current treatment.

For study participants in Part B only:

* Objective evidence of inflammation may not be required for some participants with low to moderate disease activity.
* Participants with an ASDAS score between ≥1.3 and < 2.1 (Low to Moderate Disease Activity) will require Sponsor approval prior to screening for the study, as they may not require an MRI to provide objective evidence of inflammation if on current treatment. For participants with low to moderate disease activity, MRI should only be performed if required to confirm ASAS classification.

For axSpA participants in Part B, MRI assessment of the SI joints is only required for participant eligibility criteria evaluation to assess objective inflammation in case CRP measurement at baseline is negative and the objective evidence of inflammation is required.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of dose limiting event(s) (DLE)s (Parts A and B only) | From first dose to 15 days post last dose of study drug
  To determine safety and tolerability of GRWD0715 in healthy volunteers (Part A) and participants with axSpA (Part B)
Incidence, Type and Severity of treatment related adverse events (TRAEs) | From first dose to 15 days post last dose of study drug
  To determine safety and tolerability of GRWD0715 in healthy volunteers (Part A) and participants with axSpA (Parts B and C)
Incidence, type and severity of treatment emergent adverse events (TEAEs) | From first dose to 15 days post last dose of study drug
  To determine safety and tolerability of GRWD0715 in healthy volunteers (Part A) and participants with axSpA (Parts B and C)
To determine the efficacy of GRWD0715 compared to placebo in participants with axSpA (Part D) | From baseline/Day 1 to Week 12
  Analysis of the Assessment of Spondyloarthritis International Society (ASAS) Core Outcome Set (COS). ASAS20 (improvement of 20% or more and 1 unit or more; improvement in at least 3 of 4 domains; no worsening on fourth dimension) and ASAS40 (improvement of 40% and 2 units or more; improvement in at least 3 of 4 domains; no worsening on fourth dimension) will be calculated from constituent questions with the ASAS COS clinical measures and patient reported outcomes
Analysis of SPARCC MRI activity of the SIJs (sacroiliac joints) and spine | From baseline/Day 1 to Week 12
  To determine the efficacy of GRWD0715 compared to placebo in participants with axSpA (Part D)

SECONDARY OUTCOMES:
PK Parameter Trough Concentrations | From Day 1 to Day 4 (Part A) / Day 35 (Part B) / Week 12 (Parts C and D)
  To characterise the plasma PK of GRWD0715 following single dose administration (Part A) and multiple dose administration (Parts B, C and D)
PK Parameter Cmax (Maximum observed concentration) | From Day 1 to Day 4 (Part A) / Day 35 (Part B)
  To characterise the plasma PK of GRWD0715 following single dose administration (Part A) and multiple dose administration (Part B)
PK Parameter Tmax (Time to maximum observed concentration) | From Day 1 to Day 4 (Part A) / Day 35 (Part B)
  To characterise the plasma PK of GRWD0715 following single dose administration (Part A) and multiple dose administration (Part B).
PK Parameter AUC0-t (Area under the concentration-time curve) | From Day 1 to Day 4 (Part A) / Day 35 (Part B)
  To characterise the plasma PK of GRWD0715 following single dose administration (Part A) and multiple dose administration (Parts B)
PK Parameter T1/2 (Half life) | From Day 1 to Day 4 (Part A) / Day 35 (Part B)
  To characterise the plasma PK of GRWD0715 following single dose administration (Part A) and multiple dose administration (Part B).
To assess the preliminary efficacy of GRWD0715 (Part C) | From baseline/Day 1 to Week 12
  Analysis of the Assessment of Spondyloarthritis International Society (ASAS) Core Outcome Set (COS). ASAS20 (improvement of 20% or more and 1 unit or more; improvement in at least 3 of 4 domains; no worsening on fourth dimension) and ASAS40 (improvement of 40% and 2 units or more; improvement in at least 3 of 4 domains; no worsening on fourth dimension) will be calculated from constituent questions with the ASAS COS clinical measures and patient reported outcomes
Analysis of SPARCC MRI activity of the SIJs (sacroiliac joints) and spine | From baseline/Day 1 to Week 12
  To assess the preliminary efficacy of GRWD0715 (Part C)
Incidence, Type and Severity of treatment related adverse events (TRAEs) | From first dose to 15 days post last dose of study drug
  To determine safety and tolerability of GRWD0715 in participants with axSpA (Part D).
Incidence, type and severity of treatment emergent adverse events (TEAEs) | From first dose to 15 days post last dose of study drug
  To determine safety and tolerability of GRWD0715 in participants with axSpA (Part D)

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (3):
  - University of the Sunshine Coast (UniSC), Birtinya
  - University of the Sunshine Coast (UniSC), Morayfield
  - Pioneer Clinical Research, Sydney
- Belgium (2):
  - University Ghent, Ghent
  - UZ Leuven, Leuven
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Rheumazentrum Ruhrgebiet, Ruhr-University Bochum, Bochum
- Amsterdam University Medical Center, Amsterdam, Netherlands
- Reumedika, Poznan, Poland
- University hospital Parc Tauli de Sabadell, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: No
IPD may not be shared for this Phase 1 study, or the IPD plan may be updated at a later point